CLINICAL TRIAL: NCT04761432
Title: Evaluating the Feasibility and Accuracy of a Wireless Vital Sign Monitor for Observation of Adult Patients in Uganda
Brief Title: Feasibility and Accuracy of a Wireless Vital Sign Monitor for Observation of Adult Patients in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neopenda, PBC (Industry)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MakSPH/HDREC/910
Record Dates: First submitted 2021-01-30; First posted 2021-02-18 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Critical Illness
Keywords: Critical care; Health technology; Vital sign monitoring
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Thirty (30) adult patients will be enrolled in this study. Each patient will be monitored simultaneously with the neoGuard device and a conventional patient monitor. Paired readings for temperature, respiratory rate, pulse rate and oxygen saturation will be captured every second for a maximum observation period of 1 hour.
  Interventions: Device: neoGuard

INTERVENTIONS:
Device: neoGuard — NeoGuard is a wireless wearable vital signs monitor that continuously measures temperature, pulse rate, respiratory rate and oxygen saturation.

SUMMARY:
This feasibility study will demonstrate the safety and accuracy of the Neopenda's wireless vital signs monitor, neoGuard, on 30 adult patients in a Ugandan clinical setting. The technology will be tested against a conventional patient monitor. Root mean square deviation (RMSD) and Bland-Altman plots will be used to assess concordance between paired measurements from the two equipment collected over a 1-hour period for each patient.

DETAILED DESCRIPTION:
Continuous vital sign monitoring is a basic tenet of specialized care in the developed world that is vastly underutilized in the intensive care units of most low-and-middle income countries. Despite the positive outcomes associated with vital signs monitoring (i.e. increased survival-to-discharge, lower complication rates and shorter length of hospitalization), the prohibitive costs of conventional patient monitors and the difficulty in maintaining complex medical equipment limit its accessibility in the developing world.

This feasibility study will demonstrate the safety and accuracy of the Neopenda's wireless vital signs monitor, neoGuard, on adult patients in a Ugandan clinical setting. The technology will be tested against a conventional patient monitor. Root mean square deviation (RMSD) and Bland-Altman plots will be used to assess concordance between paired measurements from the two equipment collected over a 1-hour period for each patient.

This technology innovation has large potential to impact health outcomes in low-resource settings, as it is a portable, reusable, long-lasting, cost-efficient monitoring tool designed for settings where patient loads are high and such solutions are direly needed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years (legal adult)
* Admitted for suspected or confirmed respiratory illness (excluding COVID-19)
* Stable clinical status (as determined by key physiological parameters pulse rate = 60-100 beats per minute, respiratory rate = 12-18 breaths per minute, oxygen saturation = 90 100% and temperature 36.5°C - 37.5° C)
* Willing and able to provide consent to receive vital sign monitoring

Exclusion Criteria:

* Aged <18 years
* Unstable clinical status as determined by physiological parameters (pulse rate <60 bpm, or >100bpm, respiratory rate <12 brpm or >18bpm, oxygen saturation <90%, temperature <36.5°C or >37.5°C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Accuracy limits for pulse rate, oxygen saturation, respiratory rate and temperature | 30 minutes
  Root Mean Square Deviation (RMSD) of measurements will be obtained.

SECONDARY OUTCOMES:
Feasibility success of the wireless vital sign monitor | 60 minutes
  Likert scales will be used to rate the extent to which participants agree or disagree that the neoGuard technology is appropriate and feasible in the Ugandan clinical setting. A mean feasibility score will be calculated, with a higher value indicating greater feasibility.

OTHER OUTCOMES:
Safety of the wireless vital sign monitor | 14 days
  The number of treatment-related adverse events (AE) and serious adverse events (SAE) will be categorized by their relationship to the treatment (i.e. "definitely related", "probably related", "possibly related", etc.) and severity (i.e. "mild", "moderate", "severe" or "life-threatening"). Researchers will report frequencies, descriptions and resolutions for each adverse event recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Kiwanuka, Principal Investigator — Makerere University
Locations (1):
- Jinja Regional Referral Hospital, Jinja, Uganda